CLINICAL TRIAL: NCT02262377
Title: Integrative Medicine Group Visits: A Patient-Centered Approach to Reducing Chronic Pain and Depression in a Disparate Urban Population
Brief Title: Integrative Medicine Group Visits: A Patient-Centered Approach to Reducing Chronic Pain and Depression
Acronym: IMGV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-33096
Record Dates: First submitted 2014-09-28; First posted 2014-10-13 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Chronic Pain; Depression
Keywords: Group Medical Visits; Integrative Medicine; Chronic Pain; Depression; MBSR; Mindfulness Based Stress Reduction; Web based; Virtual Patient Advocate; Internet Based
MeSH Terms: conditions — Chronic Pain; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Integrative Medicine Group Visits (Experimental): 9-week integrative medicine group visit that meets 1 time per week for 2.5 hours followed by a 3 month Web based curriculum and final group meeting
  Interventions: Behavioral: Integrative Medicine Group Visits
- Standard of Care (No Intervention): primary care visits, which include medications and advice

INTERVENTIONS:
Behavioral: Integrative Medicine Group Visits — Patients with chronic pain and depression attend group medical visits and use website and virtual patient advocate as part of the curriculum.
  Arms: Integrative Medicine Group Visits

SUMMARY:
The purpose of this study is to determine whether Integrative Medicine Group Visits (IMGV) are effective for treating patients with chronic pain and depression.

DETAILED DESCRIPTION:
The investigators propose a randomized controlled comparative effectiveness trial for patients from predominantly low-income minority backgrounds with chronic pain and depressive symptoms comparing two treatment groups: (1) A standardized, 9-session Integrative Medicine Group Visits (IMGV) protocol; (2) primary care visits including medications and provider's advice. The trial will take place at three sites: Boston Medical Center's Family Medicine Center and two affiliated federally qualified community health centers.

Patients at the three sites can self-refer or with their permission, their clinician can forward their information via email, an electronic flag or phone call to research staff. Following verbal consent, patients will be screened for eligibility by a Research Assistant either over the phone or in person. Eligible participants will then have the study explained to them by the Research Assistant and will be offered an opportunity to ask questions about the study and then invited to provide informed consent. Those participants who consent to participate will provide contact information for themselves and two additional contacts to assist with follow-up. They will then complete the baseline data survey which will consist of questionnaires on topics such as stress, pain, sleep, self-efficacy, social support, diet, exercise, relaxation, and use of pain medications. These will be administered on a tablet by a Research Assistant and should take no more than one hour to complete. Once the baseline measures have been completed, participants will be randomized to either the intervention or control condition. Once randomized, participants' clinicians will be notified via phone call, letter or email that their patient is enrolled in the study.

INTERVENTION GROUP Integrative Medicine Group Visits (IMGV)

The intervention is adapted from Mindfulness Based Stress Reduction (MBSR). For this study, those randomized to the intervention group will be asked to attend nine consecutive group visits (once a week) and a follow-up group visit at 12 weeks after the last session. During the session, a physician and co-leader facilitate each groups. Participants are taught and practice relaxation techniques at each class. The physician facilitates a discussion on health topics important to the group participants on chronic disease management, such as prevention and management of pain and associated conditions (stress re-activity, insomnia, obesity, hypertension etc.). Patients are also introduced to evidenced based complementary activities such as self-massage techniques, acupressure, and cooking classes. Finally, an optional healthy meal is served each week, creating an opportunity to model healthy nutrition and build community. Individuals randomized to IMGV will continue to receive routine medical care, including pain medications, from their primary care providers (PCPs).

Individual time spent with the group visit physician - Depending on the individual patient and his/her needs. The IMGV physician facilitator will communicate with the participants' PCPs (via electronic medical record or phone) throughout the intervention to give updates on the activities and progress of the patients.

To establish the internal validity of IMGV a research assistant will monitor the groups. An evaluation checklist of key components of the group visit will be used to assure internal validity and standardization of group IMGV curriculum across all three sites.

COMPANION WEB-BASED HOMEWORK/ HOME PRACTICE

The website serves several functions: 1) by putting all the patient materials online, it gives all patients regardless of study site the opportunity to track their health progress, participate in a monitored discussion group, and have access to audio and visual materials from class. At home, participants will complete their homework online which includes: accessing video or audio exercises or watching provider talks, which reinforce key content from the groups. 2) Our research team will use the website to track the length of time and frequency that patients practice self-care exercises at home, as well as which portions of the site the participant visits. Another component of the website is access to a Virtual Patient Advocate (VPA). The VPA will deliver a menu of mind-body activities and nutrition advice that mirrors the content of the IMGV groups.

Intervention participants will receive reminder calls each week prior to their IMGV from study staff, just as they would for other medical visits. If a participant does not attend an IMGV session, a research assistant will call to find out why they have missed the session and to remind them of the importance of attending as many sessions as possible. They will also receive letters/emails to remind them to log in to the website on a weekly basis and a letter/email to remind them about the final, follow-up session.

Control Group

Patients randomized to the control group will be given access to IMGV if desired in a non-study context at the completion of their data collection at 21 weeks (i.e., wait list control). Access to primary care providers is our control group (an approximately 15-minute usual care visit with MD, nurse practitioner (NP), physician assistant (PA) - prescribing medications, advice, standard of care recommendations).

Nine weeks after study enrollment control participants will receive a request to complete a follow-up survey which will measure the same items as the baseline survey with the exception of the demographic information and health literacy information. Finally, 21 weeks after study enrollment for the controls, participants will be asked to complete a second follow-up survey. Both follow-up surveys will be administered on a tablet by a research assistant, preferably in person, but by phone if a participant prefers.

ELIGIBILITY:
Inclusion Criteria:

* self-reported chronic pain for at least 12 weeks
* average pain intensity for the previous week >4 on a 0 to 10 numerical rating scale; PHQ-9 score >5, indicating minor depression or greater
* English fluency sufficient to follow treatment instructions and answer survey questions.

Exclusion Criteria:

* previous participation in IMGV
* new pain treatments in past month or anticipated to begin in next 3 months
* active or planned worker's compensation, disability, or personal injury claims
* known or planned pregnancy
* manic symptoms
* active suicidality
* psychotic symptoms
* no PCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Gardiner, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Upshur CC, Luckmann RS, Savageau JA. Primary care provider concerns about management of chronic pain in community clinic populations. J Gen Intern Med. 2006 Jun;21(6):652-5. doi: 10.1111/j.1525-1497.2006.00412.x. PMID 16808752
- [Background] Niazi AK, Niazi SK. Mindfulness-based stress reduction: a non-pharmacological approach for chronic illnesses. N Am J Med Sci. 2011 Jan;3(1):20-3. doi: 10.4297/najms.2011.320. PMID 22540058
- [Background] Cramer H, Lauche R, Paul A, Dobos G. Mindfulness-based stress reduction for breast cancer-a systematic review and meta-analysis. Curr Oncol. 2012 Oct;19(5):e343-52. doi: 10.3747/co.19.1016. PMID 23144582
- [Background] Cramer H, Haller H, Lauche R, Dobos G. Mindfulness-based stress reduction for low back pain. A systematic review. BMC Complement Altern Med. 2012 Sep 25;12:162. doi: 10.1186/1472-6882-12-162. PMID 23009599
- [Background] Fjorback LO, Arendt M, Ornbol E, Fink P, Walach H. Mindfulness-based stress reduction and mindfulness-based cognitive therapy: a systematic review of randomized controlled trials. Acta Psychiatr Scand. 2011 Aug;124(2):102-19. doi: 10.1111/j.1600-0447.2011.01704.x. Epub 2011 Apr 28. PMID 21534932
- [Background] Carnes D, Homer KE, Miles CL, Pincus T, Underwood M, Rahman A, Taylor SJ. Effective delivery styles and content for self-management interventions for chronic musculoskeletal pain: a systematic literature review. Clin J Pain. 2012 May;28(4):344-54. doi: 10.1097/AJP.0b013e31822ed2f3. PMID 22001667
- [Background] Eisenstat SA, Ulman K, Siegel AL, Carlson K. Diabetes group visits: integrated medical care and behavioral support to improve diabetes care and outcomes from a primary care perspective. Curr Diab Rep. 2013 Apr;13(2):177-87. doi: 10.1007/s11892-012-0349-5. PMID 23207990
- [Result] Gardiner P, Dresner D, Barnett KG, Sadikova E, Saper R. Medical group visits: a feasibility study to manage patients with chronic pain in an underserved urban clinic. Glob Adv Health Med. 2014 Jul;3(4):20-6. doi: 10.7453/gahmj.2014.011. PMID 25105072
- [Derived] Nephew BC, Incollingo Rodriguez AC, Melican V, Polcari JJ, Nippert KE, Rashkovskii M, Linnell LB, Hu R, Ruiz C, King JA, Gardiner P. Depression Predicts Chronic Pain Interference in Racially Diverse, Income-Disadvantaged Patients. Pain Med. 2022 Jul 1;23(7):1239-1248. doi: 10.1093/pm/pnab342. PMID 34908146
- [Derived] Gardiner P, Luo M, D'Amico S, Gergen-Barnett K, White LF, Saper R, Mitchell S, Liebschutz JM. Effectiveness of integrative medicine group visits in chronic pain and depressive symptoms: A randomized controlled trial. PLoS One. 2019 Dec 18;14(12):e0225540. doi: 10.1371/journal.pone.0225540. eCollection 2019. PMID 31851666
- [Derived] Gardiner P, Lestoquoy AS, Gergen-Barnett K, Penti B, White LF, Saper R, Fredman L, Stillman S, Lily Negash N, Adelstein P, Brackup I, Farrell-Riley C, Kabbara K, Laird L, Mitchell S, Bickmore T, Shamekhi A, Liebschutz JM. Design of the integrative medical group visits randomized control trial for underserved patients with chronic pain and depression. Contemp Clin Trials. 2017 Mar;54:25-35. doi: 10.1016/j.cct.2016.12.013. Epub 2016 Dec 13. PMID 27979754
- See also: Description From the Patient-Centered Outcomes Research Institute website — http://www.pcori.org/research-results/2013/integrative-medicine-group-visits-patient-centered-approach-reducing-chronic

RESULTS

PARTICIPANT FLOW:
Groups:
- Integrative Medical Group Visits: 9-week integrative medicine group visit that meets 1 time per week for 2.5 hours followed by a 3 month Web based curriculum and final group meeting
  Integrative Medicine Group Visits: Patients with chronic pain and depression attend group medical visits and use website and virtual patient advocate as part of the curriculum.
Period: Overall Study
Arm/Group | Integrative Medical Group Visits | Standard of Care
Started | 80 | 79
Completed | 68 | 73
Not Completed | 12 | 6
Not completed — Lost to Follow-up | 5 | 6
Not completed — Found ineligible after enrollment | 3 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: *We did not include intervention data on the four participants who withdrew consent.
Groups:
- Total: Total of all reporting groups
Arm/Group | Integrative Medical Group Visits | Standard of Care | Total
Number analyzed (Participants) | 76 | 79 | 155
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12.2) | 51 (12.4) | 50.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 70 | 134
  Male | 12 | 9 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 66 | 67 | 133
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 44 | 43 | 87
  White | 12 | 17 | 29
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 15 | 15 | 30
Study Sites [Count of Participants; unit: Participants]
  Boston Medical Center | 33 | 35 | 68
  Dotwell Health Center | 19 | 21 | 40
  Codman Square Health Center | 24 | 23 | 47
Income [Count of Participants; unit: Participants]
  Less than $5K | 9 | 11 | 20
  $5K-$29.99K | 36 | 41 | 77
  $30K and over | 6 | 7 | 13
  Refused/ DK/ No income | 25 | 20 | 45
Work Status [Count of Participants; unit: Participants]
  Full/ Part time | 15 | 17 | 32
  Unemployed | 10 | 12 | 22
  Retired/ Homemaker | 9 | 9 | 18
  Sick Leave/ Disability | 32 | 34 | 66
  Other | 10 | 7 | 17
Education Level [Count of Participants; unit: Participants]
  < High school/ some HS | 15 | 12 | 27
  High school degree | 22 | 31 | 53
  Some college/ AA degree | 30 | 23 | 53
  College degree or higher | 9 | 13 | 22
REALM-R score [Mean (Standard Deviation); unit: unit a scale] — Rapid Estimate of Adult Literacy in Medicine, Revised (REALM-R) is a word recognition test consisting of 11 items used to identify people at risk for poor literacy skills (Bass et al, 2003). Scores range from 0-8, and those with a score of 6 or less should be considered to be at risk for poor health literacy. You receive a point for every word pronounced properly.
  unit a scale | 6 (2.5) | 6 (2.5) | 6 (2.5)
Self Reported Substance Abuse [Count of Participants; unit: Participants]
  Current Smoker ONLY | 5 | 5 | 10
  4 or more alcoholic drinks on one occasion only | 4 | 10 | 14
  Illegal drug use only | 1 | 3 | 4
  None - smoke, drink, or use illegal drug | 35 | 34 | 69
  use at-leas 2 cigarettes or alcohol, illegal drug | 31 | 27 | 58

OUTCOME MEASURES:

1. Primary Outcome: Chronic Pain
Description: Chronic pain reflects the average scores for the severity, interference and average pain subscales from the Brief Pain Inventory (BPI) Short Form (BPI-sf). BPI-sf is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on their daily functioning on a 10 point scale from 0 to 10 where higher scores indicate higher levels of pain. Average pain was obtained by asking the participant's what their average pain was in the past 7 days. Pain interference was calculated by adding the scores for questions 8a, b, c, d, e, f, and g and then dividing by seven. Pain severity was calculated by adding the scores for questions 2, 3, 4, and 5 and then by dividing by four. The average score for each subscale was obtained by adding all respective scores and then dividing each subscale total by the total number of participants.
Time Frame: This was conducted at 21 weeks.
Population: Intention to Treat Analysis Results
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard of Care-Control: Routine primary care visits, which include medications and advice
Arm/Group | Integrative Medicine Group Visits | Standard of Care-Control
Number analyzed (Participants) | 68 | 73
units on a scale
  21 week Average pain | 6.0 (2.0) | 6.0 (2.0)
  21 week BPI Interference | 6.0 (2.7) | 5.0 (2.7)
  21 week BPI Severity | 6.0 (2.3) | 6.0 (2.0)
Statistical Analysis 1: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Intention to Treat Analysis for average chronic pain; Test type: Superiority — The ITT analysis was done for 21 week average pain; p = 0.68, Regression, Poisson — Statistical significance was set at p< 0.05; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.92 to 1.15]
Statistical Analysis 2: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority — The ITT analysis was done for 21 week BPI Interference; p = 0.36, Regression, Poisson — Statistical significance was set at p< 0.05; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.88 to 1.08]
Statistical Analysis 3: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority — The ITT analysis was done for 21 week BPI Severity; p = 0.996, Regression, Poisson — Statistical significance was set at p< 0.05; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.86 to 1.16]

2. Primary Outcome: Depression
Description: Patient Health Questionnaire (PHQ-9) measures severity of depressive symptoms. It is a sum of 9 items each with a 0-3 units on a scale. Higher scores indicate higher levels of depression. A score of 0-4 is considered minimal or none in depression severity. A score of 5-9 is considered mild in depression severity. A score of 10-14 is considered moderate in depression severity. A score of 15-19 is considered moderately severe in depression severity. A score of 20-27 is considered severe in depression severity. (Kroenke 2009) This was conducted at 21 weeks.
Time Frame: This was conducted at 21 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrative Medicine Group Visits | Standard of Care-Control
Number analyzed (Participants) | 68 | 73
units on a scale | 9.32 (5.42) | 10.15 (5.88)
Statistical Analysis 1: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority; p = 0.054, Regression, Poisson; Risk Ratio (RR) = 1.17, 95% CI 2-sided [0.99 to 1.37]

3. Primary Outcome: Pain Self Efficacy Scale
Description: Pain Self Efficacy Questionnaire (PSEQ) - used to assess the confidence in performing activities while in pain. It is the sum of 10 items each with a 0-6 scale. Scores range from 0-60 and is done by simple addition. Higher scores indicate higher levels of confidence. (Nicholas 2007) This was conducted at 21 weeks.
Time Frame: This was conducted at 21 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Integrative Medicine Group Visits | Standard of Care-Control
Number analyzed (Participants) | 68 | 73
units on a scale | 34 (14.7) | 38 (13.5)
Statistical Analysis 1: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority; p = 0.98, Regression, Poisson; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.89 to 1.13]

4. Primary Outcome: Pain Medication Use
Description: Number of participants reported pain medication in the past seven day. This was obtained at 21 weeks.
Time Frame: This was conducted at 21 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Integrative Medicine Group Visits | Standard of Care-Control
Number analyzed (Participants) | 68 | 73
Participants | 49 | 60
Statistical Analysis 1: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority; Odds Ratio; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.18 to 0.98]

5. Secondary Outcome: Emergency Department Use
Description: Number of emergency room visits based on chart review data collection.
Time Frame: This was collected at 21 weeks.
Measure: Number; unit: participants
Arm/Group | Integrative Medicine Group Visits | Standard of Care-Control
Number analyzed (Participants) | 68 | 73
participants | 9 | 9
Statistical Analysis 1: Comparison: Integrative Medicine Group Visits vs Standard of Care-Control; Test type: Superiority; Odds Ratio; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.90 to 1.14]

ADVERSE EVENTS:
Groups:
- All Participants: All participants included in the RCT.
Arm/Group | Integrative Medical Group Visits | Standard of Care | All Participants
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/79 | 0/155
Serious Adverse Events (participants affected / at risk) | 1/76 | 1/79 | 2/155
Other Adverse Events (participants affected / at risk) | 19/76 | 13/79 | 32/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrative Medical Group Visits (N=76) | Standard of Care (N=79) | All Participants (N=155)
Hospitalization unrelated to study (General disorders) | 1 (1) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Integrative Medical Group Visits (N=76) | Standard of Care (N=79) | All Participants (N=155)
Non Serious Adverse Events (General disorders) | 19 (22) | 13 (20) | 32 (42) — Muscle Strain, pain in new location, ER visits, fell off chair, falling down, other.These adverse event terms cannot be separated.

LIMITATIONS AND CAVEATS:
Our limitations for this study includes: study participation (intervention group did not all attend IMGV and not everyone in control group attended PCP visit), no data on baseline antidepressants medication, only English speaking patients included.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No